CLINICAL TRIAL: NCT04401046
Title: COVID-19 EPIDEMIC Reorganisation of Cancer Patient Care: Self- Evaluation of Potential Post-traumatic Stress Disorder
Brief Title: COVID-19 and Reorganisation of Cancer Patient Care: Self- Evaluation of Potential Post-traumatic Stress Disorder
Acronym: COVID-TRAUMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: COVID-TRAUMA-IPC 2020-026
Record Dates: First submitted 2020-05-22; First posted 2020-05-26 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Cancer
Keywords: COVID-19; POST TRAUMATIC STRESS; CANCER; ANXIETY; REORGANISATION OF CARE
MeSH Terms: conditions — Neoplasms; COVID-19; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post traumatic stress and anxiety evaluation (Experimental)
  Interventions: Other: Survey to assess Post traumatic stress and anxiety at inclusion and 6 months later

INTERVENTIONS:
Other: Survey to assess Post traumatic stress and anxiety at inclusion and 6 months later — The first survey will include questions relative to sociodemographic characteristics, existence of psychological troubles; living conditions in the Covid19 pandemic context; IES-R, Stait Trait Anxiety, and the fear of a cancer recurrence scales, satisfaction with cancer care and medical status of patients (diagnosis, ongoing treatment, follow-up of the disease).

SUMMARY:
The COVID-19 pandemic is a traumatic event which could lead to a greater risk of developing post-traumatic stress disorder, especially in cancer patients who feel more at risk of contracting the virus, and fear developing serious symptoms. The study's primary objective is to measure the presence of a potential post-traumatic stress disorder in cancer patients, and to assess the associated factors. The secondary objectives are to measure patients' anxiety, as well as their perception of both the management of their cancer care, and their fear of a cancer recurrence.

It is a prospective, multi-centric study using self-assessing survey offered to cancer patients currently under ongoing care or treatment. The surveys will be sent by post at the beginning of the study, and again 6 months later. Expecting a participation rate of 40%, 4000 patients will be contacted, over a period of 3 months, in order to receive 1600 responses, and 640 responses 6 months later.

Researching the factors associated with the appearance of post-traumatic stress could lead to better screening of patient disorders in highly anxiety-provoking crisis situations. As a result, it would lead to an improvement of their care, healthcare organization, and their follow-up in the case of a new epidemic or any other stressful event of this magnitude. Furthermore, promoting the patient's expression capabilities favors their implication in their care, and facilitates the development of health democracy.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman, age>18
* Diagnosis of cancer (solid tumor or hematology)
* Out patient or patient Under surveillance

Exclusion Criteria:

* Refusal to participate in the study
* Emergency, person deprived of liberty
* hospitalized patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1096 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-11-26 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Score of the Impact of Event Scale Revisited scale | at inclusion and 6 months later

SECONDARY OUTCOMES:
Factors associated with post-traumatic stress disorder | at inclusion and 6 months later
  The factors associated with post traumatic stress, measured by the Impact of Event Scale Revisited scale
Measure of the patient's anxiety | at inclusion and 6 months later
  The measure of anxiety, measured by the State-Trait Anxiety Questionnaire
proportion of patients perceiving poorer management of their cancer care since the start of the COVID-19 epidemic. | at inclusion and 6 months later
proportion of patients perceiving the implementation of all necessary measures to reduce the risk of exposure to COVID-19 | at inclusion and 6 months later
proportion of patients stating that remote consultation is as useful as a face-to-face consultation | at inclusion and 6 months later
proportion of patients with access to a clinical psychology consultation (at the hospital or on the phone) | at inclusion and 6 months later
Score on the cancer recurrence scale | at inclusion and 6 months later

CONTACTS AND LOCATIONS:
Overall Officials: Gwenaelle GRAVIS, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli-Calmettes, Marseille, France